CLINICAL TRIAL: NCT02014402
Title: A Prospective, Randomized, Double-blind, Phase II Study to Evaluate the Safety and Efficacy of Topical Thrombin (Human) Grifols as an Adjunct to Hemostasis During Vascular, Hepatic, Soft Tissue, and Spinal Open Surgeries
Brief Title: Safety and Efficacy of Topical Thrombin (Human) Grifols as an Adjunct to Hemostasis During Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IG1202 (IG1202-A, -B, -C, -D)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Hemostasis
Keywords: Vascular surgery; Hepatic surgery; Soft tissue surgery; Spinal surgery
MeSH Terms: interventions — Thrombin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IG1202-A (Vascular) (Experimental)
  Interventions: Biological: Human thrombin; Biological: Bovine thrombin
- IG1202-B (Hepatic) (Experimental)
  Interventions: Biological: Human thrombin; Biological: Bovine thrombin
- IG1202-C (Soft Tissue) (Experimental)
  Interventions: Biological: Human thrombin; Biological: Bovine thrombin
- IG1202-D (Spinal) (Experimental)
  Interventions: Biological: Human thrombin; Biological: Bovine thrombin

INTERVENTIONS:
Biological: Human thrombin — Thrombin purified from human plasma reconstituted as a 1000 IU/mL solution in blinded syringes and applied using Gelfoam® sponges
Biological: Bovine thrombin — Thrombin of bovine origin reconstituted as a 1000 IU/mL solution in blinded syringes and applied using Gelfoam® sponges

SUMMARY:
This purpose of this clinical trial was to study the safety and efficacy of Topical Thrombin (Human) Grifols as an add-on treatment to help stop bleeding during vascular, liver, soft tissue, and spinal surgical procedures.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blind, controlled, Phase II study to evaluate the safety and efficacy of Topical Thrombin (Human) Grifols as an adjunct to hemostasis during vascular (IG1202-A), hepatic (IG1202-B), soft tissue (IG1202-C), and spinal (IG1202-D) surgical procedures. Approximately 180 subjects were randomized into 1 of 2 treatment groups in a 2:1 ratio: Topical Thrombin (Human) Grifols (120 subjects) or Bovine Thrombin JMI (60 subjects) among the 4 types of surgeries. Randomized subjects were evaluated for identification of a target bleeding site (TBS) in which control of bleeding by conventional surgical techniques (including suture, ligature and cautery) was ineffective or impractical and required an adjunct treatment to achieve hemostasis. The Investigator rated the intensity of bleeding at the TBS. Topical Thrombin (Human) Grifols or Bovine Thrombin JMI was applied to the TBS and the time to hemostasis was assessed at various timepoints during a 5-minute observation period.

Subjects were evaluated by surgery type and by integrated analysis of clinical studies IG1202-A, IG1202-B, IG1202-C, and IG1202-D.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative (at Baseline Assessments Visit) hemoglobin (Hgb) ≥9.0 g/dL (deciliter)
* Pre-operative (at Baseline Assessments Visit) fibrinogen level ≥150 mg/dL (functional method).
* Required one of the following procedures:

  1. An elective (non-emergency), open (non-laparoscopic; non- endovascular) surgical procedure involving a native artery-graft end-to-side proximal anastomosis utilizing coated or uncoated polytetrafluoroethylene (PTFE) graft (IG1202-A).
  2. An elective (non-emergency), open (non-laparoscopic) hepatic resection (anatomic and non-anatomic resections of at least one anatomical hepatic segment or equivalent tissue volume) (IG-1202-B).
  3. An elective (non-emergency), open (non-laparoscopic), surgical procedure involving soft (non-parenchymous) tissue (IG1202-C).
  4. An elective (non-emergency), spinal surgical procedure in which the epidural venous plexus was exposed (IG1202-D).
* A target bleeding site (TBS) was identified according to the Investigator's judgment, and the TBS had mild or moderate bleeding according to the Investigator's judgment.

Exclusion Criteria:

* Required surgical procedure due to trauma (except for spinal surgery).
* Infection in the anatomic surgical area.
* History of severe (e.g. anaphylactic) reactions to blood or to any blood-derived (human or animal) product.
* Previous known sensitivity to any Topical Thrombin (Human) Grifols component, any Bovine Thrombin JMI component, porcine collagen, and heparin or protamine (vascular surgery only) component.
* Received an organ transplant.
* Underwent another concurrent major surgical intervention beyond the liver (applied to hepatic surgery [IG1202-B] only; concurrent interventions on the pancreas, gall bladder, bile duct, or intestines were allowed).
* Underwent a re-operative procedure, which was defined as a second, or successive, surgical procedure on the same anatomic location.
* Underwent other vascular procedures during the same surgical session (applied to vascular surgery [IG1202-A] only; stenting and/or endarterectomy of the same artery were allowed).
* Underwent a therapeutic surgical procedure within 30 days from screening (diagnostic procedures were allowed).
* Previously included in this trial (i.e. each subject could only be enrolled once in this study).
* TBS could not be identified according to the investigator's judgment.
* TBS had a severe bleeding according to the Investigator's judgment.
* Occurrence of major intra-operative complications that required resuscitation or deviation from the planned surgical procedure.
* Application of any topical haemostatic material on the resection surface of the liver prior to application of the study treatment (applied to hepatic surgery [IG1202-B] only).
* Radiofrequency precoagulation of the liver resection surface, except focal use of radiofrequency as primary haemostatic treatment (applied to hepatic surgery [IG1202-B] only).
* Intra-operative change in planned surgical procedure which resulted in subject no longer meeting preoperative inclusion and/or exclusion criteria.
* Application of any topical haemostatic material on the cut soft tissue surface prior to application of the study treatment (applied to soft tissue surgery [IG1202-C] only).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - 805, Tucson, Arizona
  - 602, Los Angeles, California
  - 700, 801, Pasadena, California
  - 803, Boulder, Colorado
  - 908, Hartford, Connecticut
  - 601, Washington D.C., District of Columbia
  - 507, Gainesville, Florida
  - 501, 901, Jacksonville, Florida
  - 604, Evanston, Illinois
  - 804, Lexington, Kentucky
  - 905, Baltimore, Maryland
  - 902, Jackson, Mississippi
  - 800, Las Vegas, Nevada
  - 600, New York, New York
  - 606, Poughkeepsie, New York
  - 508, Chapel Hill, North Carolina
  - 503, Fort Worth, Texas
  - 900, Houston, Texas
  - 605, Salt Lake City, Utah
  - 802, Spokane, Washington

REFERENCES:
- [Derived] Minkowitz H, Navarro-Puerto J, Lakshman S, Singla S, Cousar C, Kim R, Villavicencio A, Kirksey L, Ayguasanosa J; Clinical Investigation Study Group on Topical Thrombin (Human) Grifols in Surgery. Prospective, Randomized, Phase II, Non-Inferiority Study to Evaluate the Safety and Efficacy of Topical Thrombin (Human) Grifols as Adjunct to Hemostasis During Vascular, Hepatic, Soft Tissue, and Spinal Open Surgery. J Am Coll Surg. 2019 Nov;229(5):497-507.e1. doi: 10.1016/j.jamcollsurg.2019.07.008. Epub 2019 Jul 31. PMID 31376435

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IG1202-A (Vascular) | IG1202-B (Hepatic) | IG1202-C (Soft Tissue) | IG1202-D (Spinal)
Started | 31 | 30 | 35 | 85
Human Thrombin | 20 | 20 | 23 | 57
Bovine Thrombin | 11 | 10 | 12 | 28
Completed | 29 | 27 | 32 | 82
Not Completed | 2 | 3 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 1
Not completed — Subject did not have transportation | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IG1202-A (Vascular) | IG1202-B (Hepatic) | IG1202-C (Soft Tissue) | IG1202-D (Spinal) | Total
Number analyzed (Participants) | 31 | 30 | 35 | 85 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age categories are provided by number of subjects in the Human Thrombin and Bovine Thrombin treatment groups
  years
    Human Thrombin: number analyzed (Participants) | 20 | 20 | 23 | 57 | 120
    Human Thrombin | 66.30 (12.427) | 57.50 (13.987) | 47.52 (13.885) | 54.32 (16.733) | 55.54 (16.017)
    Bovine Thrombin: number analyzed (Participants) | 11 | 10 | 12 | 28 | 61
    Bovine Thrombin | 71.82 (9.857) | 56.50 (14.455) | 47.67 (12.434) | 54.04 (17.240) | 56.39 (16.464)
Age, Customized [Count of Participants; unit: Participants] — Population: Age categories are provided by number of subjects in the Human Thrombin and Bovine Thrombin treatment groups
  Participants
    12-17: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
    12-17: Human Thrombin | 0 | 0 | 0 | 1 | 1
    12-17: Bovine Thrombin | 0 | 0 | 0 | 1 | 1
    18-64: number analyzed (Participants) | 12 | 21 | 31 | 59 | 123
    18-64: Human Thrombin | 9 | 13 | 20 | 40 | 82
    18-64: Bovine Thrombin | 3 | 8 | 11 | 19 | 41
    >=65: number analyzed (Participants) | 19 | 9 | 4 | 24 | 56
    >=65: Human Thrombin | 11 | 7 | 3 | 16 | 37
    >=65: Bovine Thrombin | 8 | 2 | 1 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender categories are provided by number of subjects in the Human Thrombin and Bovine Thrombin treatment groups
  Participants
    Human Thrombin: number analyzed (Participants) | 20 | 20 | 23 | 57 | 120
    Human Thrombin: Female | 8 | 10 | 23 | 29 | 70
    Human Thrombin: Male | 12 | 10 | 0 | 28 | 50
    Bovine Thrombin: number analyzed (Participants) | 11 | 10 | 12 | 28 | 61
    Bovine Thrombin: Female | 4 | 9 | 11 | 18 | 42
    Bovine Thrombin: Male | 7 | 1 | 1 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race categories are provided by number of subjects in the Human Thrombin and Bovine Thrombin treatment groups
  Participants
    White (Caucasian): number analyzed (Participants) | 23 | 19 | 23 | 82 | 147
    White (Caucasian): Human Thrombin | 14 | 13 | 15 | 55 | 97
    White (Caucasian): Bovine Thrombin | 9 | 6 | 8 | 27 | 50
    Black or African American: number analyzed (Participants) | 8 | 6 | 10 | 2 | 26
    Black or African American: Human Thrombin | 6 | 5 | 6 | 2 | 19
    Black or African American: Bovine Thrombin | 2 | 1 | 4 | 0 | 7
    Asian: number analyzed (Participants) | 0 | 2 | 2 | 0 | 4
    Asian: Human Thrombin | 0 | 0 | 2 | 0 | 2
    Asian: Bovine Thrombin | 0 | 2 | 0 | 0 | 2
    American Indian or Alaskan Native: number analyzed (Participants) | 0 | 1 | 0 | 1 | 2
    American Indian or Alaskan Native: Human Thrombin | 0 | 1 | 0 | 0 | 1
    American Indian or Alaskan Native: Bovine Thrombin | 0 | 0 | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander: Human Thrombin | 0 | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander: Bovine Thrombin | 0 | 0 | 0 | 0 | 0
    Other: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
    Other: Human Thrombin | 0 | 0 | 0 | 0 | 0
    Other: Bovine Thrombin | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Hemostasis by Five Minutes After Treatment Start at the TBS
Description: Subjects achieving hemostasis at the target bleeding site by 5 minutes following the start of treatment without the occurrence of re-bleeding until the completion of surgical closure
Time Frame: From start of treatment until 5 minutes after treatment start
Population: Data are presented for subjects in the Human Thrombin and Bovine Thrombin treatment groups in the modified intent-to-treat (mITT) population
Measure: Number; unit: percent of subjects achieving hemostasis
Groups:
- Overall (IG1202-A, IG1202-B, IG1202-C, and IG1202-D): Human thrombin: Thrombin purified from human plasma reconstituted as a 1000 IU/mL solution in blinded syringes and applied using Gelfoam® sponges
  Bovine thrombin: Thrombin of bovine origin reconstituted as a 1000 IU/mL solution in blinded syringes and applied using Gelfoam® sponges
Arm/Group | IG1202-A (Vascular) | IG1202-B (Hepatic) | IG1202-C (Soft Tissue) | IG1202-D (Spinal) | Overall (IG1202-A, IG1202-B, IG1202-C, and IG1202-D)
Number analyzed (Participants) | 31 | 30 | 35 | 85 | 181
percent of subjects achieving hemostasis
  Human Thrombin: number analyzed (Participants) | 20 | 20 | 23 | 57 | 120
  Human Thrombin | 75.0 | 75.0 | 73.9 | 82.5 | 78.3
  Bovine Thrombin: number analyzed (Participants) | 11 | 10 | 12 | 28 | 61
  Bovine Thrombin | 54.5 | 80.0 | 91.7 | 85.7 | 80.3

2. Secondary Outcome: Cumulative Proportion of Subjects Having Achieved Hemostasis at the Target Bleeding Site by Specified Time Points
Description: Cumulative proportion of subjects having achieved hemostasis by each of the following time points:
  * At 3 minutes following start of study treatment
  * At 4 minutes following start of study treatment
Time Frame: From start of treatment until 4 minutes after treatment start
Population: Data are presented for subjects in the Human Thrombin and Bovine Thrombin treatment groups in the mITT population
Measure: Number; unit: percent of subjects achieving hemostasis
Arm/Group | IG1202-A (Vascular) | IG1202-B (Hepatic) | IG1202-C (Soft Tissue) | IG1202-D (Spinal) | Overall (IG1202-A, IG1202-B, IG1202-C, and IG1202-D)
Number analyzed (Participants) | 31 | 30 | 35 | 85 | 181
percent of subjects achieving hemostasis
  Hemostasis by 3 minutes: Human Thrombin: number analyzed (Participants) | 20 | 20 | 23 | 57 | 120
  Hemostasis by 3 minutes: Human Thrombin | 40.0 | 45.0 | 73.9 | 70.2 | 61.7
  Hemostasis by 3 minutes: Bovine Thrombin: number analyzed (Participants) | 11 | 10 | 12 | 28 | 61
  Hemostasis by 3 minutes: Bovine Thrombin | 36.4 | 60.0 | 75.0 | 71.4 | 63.9
  Hemostasis by 4 minutes: Human Thrombin: number analyzed (Participants) | 20 | 20 | 23 | 57 | 120
  Hemostasis by 4 minutes: Human Thrombin | 50.0 | 65.0 | 73.9 | 78.9 | 70.8
  Hemostasis by 4 minutes: Bovine Thrombin: number analyzed (Participants) | 11 | 10 | 12 | 28 | 61
  Hemostasis by 4 minutes: Bovine Thrombin | 45.5 | 70.0 | 91.7 | 78.6 | 73.8

3. Secondary Outcome: Prevalence of Treatment Failures
Description: Protocol-defined bleeding at the target bleeding site after the start of treatment or the use of alternative hemostatic treatments or maneuvers at the target bleeding site after the start of treatment
Time Frame: From start of treatment up to surgical closure by layers of the exposed surgical field containing the TBS, a median of 34 minutes
Population: Data are presented for subjects in the Human Thrombin and Bovine Thrombin treatment groups in the mITT population
Measure: Number; unit: percent of subjects
Arm/Group | IG1202-A (Vascular) | IG1202-B (Hepatic) | IG1202-C (Soft Tissue) | IG1202-D (Spinal) | Overall (IG1202-A, IG1202-B, IG1202-C, and IG1202-D)
Number analyzed (Participants) | 31 | 30 | 35 | 85 | 181
percent of subjects
  Human Thrombin: number analyzed (Participants) | 20 | 20 | 23 | 57 | 120
  Human Thrombin | 25.0 | 25.0 | 26.1 | 17.5 | 21.7
  Bovine Thrombin: number analyzed (Participants) | 11 | 10 | 12 | 28 | 61
  Bovine Thrombin | 45.5 | 20.0 | 8.3 | 14.3 | 19.7

ADVERSE EVENTS:
Time Frame: Adverse event data (safety population) were collected from the time informed consent was obtained through the Post-Operative Day 30
Groups:
- IG1202-A (Vascular): Human Thrombin; IG1202-B (Hepatic): Human Thrombin; IG1202-C (Soft Tissue): Human Thrombin; IG1202-D (Spinal): Human Thrombin; Overall (IG1202-A, -B, -C, and -D): Human Thrombin: Human thrombin: Thrombin purified from human plasma reconstituted as a 1000 IU/mL solution in blinded syringes and applied using Gelfoam® sponges
- IG1202-A (Vascular): Bovine Thrombin; IG1202-B (Hepatic): Bovine Thrombin; IG1202-C (Soft Tissue): Bovine Thrombin; IG1202-D (Spinal): Bovine Thrombin; Overall (IG1202-A, -B, -C, and -D): Bovine Thrombin: Bovine thrombin: Thrombin of bovine origin reconstituted as a 1000 IU/mL solution in blinded syringes and applied using Gelfoam® sponges
Arm/Group | IG1202-A (Vascular): Human Thrombin | IG1202-A (Vascular): Bovine Thrombin | IG1202-B (Hepatic): Human Thrombin | IG1202-B (Hepatic): Bovine Thrombin | IG1202-C (Soft Tissue): Human Thrombin | IG1202-C (Soft Tissue): Bovine Thrombin | IG1202-D (Spinal): Human Thrombin | IG1202-D (Spinal): Bovine Thrombin | Overall (IG1202-A, -B, -C, and -D): Human Thrombin | Overall (IG1202-A, -B, -C, and -D): Bovine Thrombin
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/11 | 0/20 | 0/10 | 0/23 | 0/12 | 0/57 | 1/28 | 0/120 | 2/61
Serious Adverse Events (participants affected / at risk) | 3/20 | 2/11 | 2/20 | 1/10 | 1/23 | 0/12 | 4/57 | 3/28 | 10/120 | 6/61
Other Adverse Events (participants affected / at risk) | 12/20 | 7/11 | 20/20 | 9/10 | 23/23 | 12/12 | 49/57 | 24/28 | 104/120 | 52/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IG1202-A (Vascular): Human Thrombin (N=20) | IG1202-A (Vascular): Bovine Thrombin (N=11) | IG1202-B (Hepatic): Human Thrombin (N=20) | IG1202-B (Hepatic): Bovine Thrombin (N=10) | IG1202-C (Soft Tissue): Human Thrombin (N=23) | IG1202-C (Soft Tissue): Bovine Thrombin (N=12) | IG1202-D (Spinal): Human Thrombin (N=57) | IG1202-D (Spinal): Bovine Thrombin (N=28) | Overall (IG1202-A, -B, -C, and -D): Human Thrombin (N=120) | Overall (IG1202-A, -B, -C, and -D): Bovine Thrombin (N=61)
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dural tear (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IG1202-A (Vascular): Human Thrombin (N=20) | IG1202-A (Vascular): Bovine Thrombin (N=11) | IG1202-B (Hepatic): Human Thrombin (N=20) | IG1202-B (Hepatic): Bovine Thrombin (N=10) | IG1202-C (Soft Tissue): Human Thrombin (N=23) | IG1202-C (Soft Tissue): Bovine Thrombin (N=12) | IG1202-D (Spinal): Human Thrombin (N=57) | IG1202-D (Spinal): Bovine Thrombin (N=28) | Overall (IG1202-A, -B, -C, and -D): Human Thrombin (N=120) | Overall (IG1202-A, -B, -C, and -D): Bovine Thrombin (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 2 | 0 | 4 | 3
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 4 | 2 | 1 | 7 | 3 | 12 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 8 | 6 | 10 | 4 | 13 | 6 | 33 | 16
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 6 | 2 | 2 | 2 | 2 | 6 | 10
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 4 | 3
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 4 | 2
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 5 | 3 | 7 | 5 | 22 | 11 | 33 | 19 | 67 | 38
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intra-abdominal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 3 | 1 | 0 | 6 | 2 | 12 | 4
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 4 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 0 | 1 | 1 | 0 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 5 | 1 | 0 | 2 | 1 | 2 | 6 | 5
Visceral pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 4 | 2
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Urine output decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 10 | 5 | 11 | 6
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 3 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 9 | 3 | 11 | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the study, after providing Sponsor 30 days' notice prior to submitting a manuscript or other materials related to the study to any outside party. At Sponsor's request, site will remove any confidential information (other than study results) and site will, upon Sponsor's request, delay publication or presentation for a period of up to 120 days to allow Sponsor to protect its interests in any Sponsor interventions.